CLINICAL TRIAL: NCT04777604
Title: Development of a Prediction Platform for Neoadjuvant Treatment and Prognosis in Pancreatic Cancer Using Ex Vivo Analysis of Organoid Culture
Brief Title: Development of a Prediction Platform for Neoadjuvant Treatment and Prognosis in Pancreatic Cancer Using Organoid
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, JooKyung Park, Associate Professor, Samsung Medical Center
Other Study IDs: 2020-12-106
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with resectable pancreatic cancer after neoadjuvant chemotherapy
  Interventions: Other: Organoid

INTERVENTIONS:
Other: Organoid — The investigators create organoid from the pancreatic cancer tissue obtained via EUS-FNA and EUS-FNB within the pancreatic cancer diagnostic process. And also the investigators create organoid from the pancreatic cancer tissue obtained after surgery as part of the pancreatic cancer treatment process. Check for the reactivity to anti-cancer drugs through cell viability assay after treating with various anti-cancer drugs, such as anti-cancer drugs used as neoadjuvant chemotherapy for pancreatic cancer to the organoid. Also, perform genomic analysis on each organoid, and then check if there are any unique genomic mutations for each organoid. By recognizing the relationship between the unique genomic mutations and reactivity to the anti-cancer drug within patients with resectable pancreatic cancer after neoadjuvant chemotherapy, the investigators aim to strategize appropriate neoadjuvant chemotherapy before surgery, thus developing a platform to predict the outcomes of each patient.

SUMMARY:
The investigators create organoid from the pancreatic cancer tissue obtained via EUS-FNA and EUS-FNB within the pancreatic cancer diagnostic process. And also the investigators create organoid from the pancreatic cancer tissue obtained after surgery as part of the pancreatic cancer treatment process. Check for the reactivity to anti-cancer drugs through cell viability assay after treating with various anti-cancer drugs, such as anti-cancer drugs used as neoadjuvant chemotherapy for pancreatic cancer to the organoid. Also, perform genomic analysis on each organoid, and then check if there are any unique genomic mutations for each organoid. By recognizing the relationship between the unique genomic mutations and reactivity to the anti-cancer drug within pancreatic cancer patients eligible for surgery, the investigators aim to strategize appropriate neoadjuvant chemotherapy before surgery, thus developing a platform to predict the outcomes of each patient.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old or older
2. Newly discovered pancreatic cancer and not a relapse
3. Diagnosed with pancreatic cancer via EUS-FNA, EUS-FNB before surgery
4. who is in need of neoadjuvant chemotherapy before surgery
5. Patients who can undergo surgery for pancreatic cancer after neoadjuvant chemotherapy
6. Diagnosed with pancreatic cancer from the final tissue pathology diagnosis after surgery
7. Able to make decisions for oneself for participation
8. Has obtained voluntary consent in written form (if 70 years of age or older, receive consent from the guardian as well)

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A patient who is in need of neoadjuvant chemotherapy before surgery, having been diagnosed with pancreatic cancer via EUS-FNA and EUS-FNB at Samsung Medical Center. And a patient who is eligible for surgery after neoadjuvantchemotherapy.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2025-01-07 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | From date of initiation of adjuvant chemotherapy after surgery until the date of death from any cause, assessed up to 36 months
  The percentage of people in a group who are still alive for a certain period of time after they were started adjuvant chemotherapy for pancreatic cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No